CLINICAL TRIAL: NCT03831516
Title: Non-Invasive 3D Mapping for Identifying Origin and Preferential Propagation of Ventricular Arrhythmias
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Stavros E Mountantonakis, Associate Director of Cardiac Electrophysiology, Northwell Health
Other Study IDs: 18-0364
Record Dates: First submitted 2019-01-25; First posted 2019-02-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Premature Ventricular Complex; Ventricular Arrythmia
Keywords: Ablation; Ventricular Tachycardia; Mapping
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Non Invasive Electroanatomical Mapping: Patients will undergo non invasive electroanatomical mapping (CardioInsight by Medtronic) prior and during an invasive electrophysiology study and ablation of ventricular Arrhythmias.
  Interventions: Diagnostic Test: Non Invasive Electroanatomical Mapping

INTERVENTIONS:
Diagnostic Test: Non Invasive Electroanatomical Mapping — All patients will undergo non contrast CT chest and be fitted with the Medtronic CardioInsight wearable 252 electrode vest. Non invasive electroanatomical maps of the ventricular arrhythmia will be created. All patients will be then brought to the electrophysiology laboratory and undergo an invasive electrophysiology study and ablation of the ventricular arrhythmia.

SUMMARY:
This study will measure the diagnostic sensitivity and specificity of the Medtronic CardioInsight wearable 252 electrode vest in predicting the chamber of origin of premature ventricular complexes (PVCs) and compare its diagnostic accuracy with the standard 12- lead ECG.

DETAILED DESCRIPTION:
Until recently, the only non-invasive diagnostic modality to help identify the location of ventricular arrhythmias was the 12 lead ECG. The Medtronic CardioInsight wearable vest is a recently FDA approved diagnostic modality noninvasive, single beat cardiac mapping system that provides 3D electroanatomic maps of the ventricular chambers. CardioInsight projects unipolar signals collected from a 252-electrode vest to cardiac chambers imaged with a non-contrast CT of the chest. The created non-invasive 3D electroanatomical maps can be evaluated by the physicians pre-procedurally but also during the actual electrophysiology study (EPS).

The technology has been approved by FDA for non-invasive mapping of any arrhythmias, however there is little evidence on its value in predicting the origin of ventricular arrhythmias and its proven diagnostic superiority over the standard 12-lead ECG.

With this study the investigators seek to assess the sensitivity and specificity of CardioInsight in predicting the chamber of origin of ventricular arrhythmias and compare its diagnostic accuracy with the standard 12-lead ECG. The study will include thirty patients with ventricular arrhythmias undergoing EPS and ablation. The day of the procedure patients will be fitted with the CardioInsight vest and undergo a non-contrast CT chest. Spontaneous arrhythmias will be recorded and noninvasive 3D maps will be created prior and during the EPS. The non-invasive maps will be used, per operator discretion, in designing mapping and ablative strategies during the EPS. The true origin of the arrhythmia will be determined during the EPS. In addition, the investigators will perform threshold pacing from common site of idiopathic ventricular arrhythmias. The 12-lead ECGs and non-invasive maps will be stored for off line review and analysis.

Non-invasive maps, as well as ECGs of spontaneous arrhythmias and pacemaps will be evaluated off line by 2 electrophysiologists blinded to the results of the EPS. The sensitivity and specificity of the 12 lead ECG, as well as the non-invasive maps, in predicting the site of origin of the ventricular arrhythmias and pacemaps will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PVCs or VT requiring EPS for:
* Symptomatic arrhythmias
* High PVC burden
* Presence of cardiomyopathy
* Risk stratification to determine which patients to offer ablative vs medical therapy and for ICD implantation if deemed high risk for sudden cardiac death.

Exclusion Criteria:

* Patients in acute coronary syndrome
* Patient with congestive heart failure in acute decompensation
* Patients in rapid atrial fibrillation
* Patients requiring persistent ventricular pacing
* Patient who refuse to undergo EPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ventricular arrhythmias (premature ventricular complexes - PVC or ventricular tachycardias - VT) requiring EPS for risk stratification or ablation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Predicting Origin | 12 month
  Measure the diagnostic sensitivity and specificity of non-invasive mapping system in predicting origin of spontaneous ventricular arrhythmias in patients undergoing EPS

SECONDARY OUTCOMES:
Preferential Electrical Propagation of Ventricular Arrhythmia | 12 month
  Identify and describe the presence of preferential electrical propagation of ventricular arrhythmias in patients undergoing EPS.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Mountantonakis, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No